CLINICAL TRIAL: NCT06946056
Title: Evaluation of the Effect of Biofiller PRP Application on Range of Motion, Pain, Quality of Life and Femoral Cartilage Thickness in Knee Osteoarthritis
Brief Title: Evaluation of the Effect of Biofiller PRP Application on Knee Osteoarthritis
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Necmettin Erbakan University (Other)
Responsible Party: Principal Investigator, Banu Ordahan, professor, Necmettin Erbakan University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Büşra Demirtaş
Record Dates: First submitted 2025-04-09; First posted 2025-04-27 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Knee Osteoarthritis; Biofiller PRP; Femoral Cartilage Thickness
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Biofiller platelet rich plasma (Active Comparator): Ten ml of the patient's blood wasdrawn in a syringe pre-filled with 1 mLacid citrate dextrose(anticoagulant). It wascentrifuged firstat 4000 rotations per minute (RPM)for 15 min and thenat 1500 RPM for 5 min. The upper part,i.e.,platelet-poor plasma (PPP) was withdrawn in a 5 mL syringe. PRP was incubated in hot incubator at 100a °C for 5 min and then cooled in a refrigerator for 5 min.
  Interventions: Other: biofiller prp
- Platelet rich plasma (Active Comparator): Ten ml of the patient's blood wasdrawn in a syringe pre-filled with 1 mLacid citrate dextrose(anticoagulant). It wascentrifuged firstat 4000 rotations per minute (RPM)for 15 min and thenat 1500 RPM for 5 min. The upper part,i.e.,platelet-poor plasma (PPP) was withdrawn in a 5 mL syringe
  Interventions: Other: biofiller prp

INTERVENTIONS:
Other: biofiller prp — Ten ml of the patient's blood was drawn in a syringe pre-filled with 1 mLacid citrate dextrose(anticoagulant). It wascentrifuged firstat 3500 rotations per minute (RPM)for 15 min and thenat 1500 RPM for 5 min. The upper part,i.e.,platelet-poor plasma (PPP) waswithdrawn in a 5 mL syringe. PPP wasincubated in hot water at 100a °C for 5 min and then cooled in a refrigerator for 5 min.The PRP injection was performed in a standardized manner and injected into the IA surface of the affected knee joint

SUMMARY:
The aim of this study is to evaluate the effects of biofiller PRP, on pain, range of motion, quality of life, and femoral cartilage thickness in patients with knee osteoarthritis.

DETAILED DESCRIPTION:
Patients who are admitted and diagnosed with knee osteoarthritis based on anamnesis, physical examination and imaging methods are included in the study

ELIGIBILITY:
Inclusion Criteria:

1-45-65 years old 2-Diagnosis of knee OA according to ACR clinical and radiological diagnostic criteria 3-Kellgren Lawrence stage II or III 4-Knee pain for at least 6 months 5-Visual analog scale (VAS) score of at least 3 or more

Exclusion Criteria:

1 - History of surgery or traumatic injury 2-Inflammatory arthritis 3-History of cancer, bleeding diathesis and psychiatric disease 4-Those who have a disease that limits their participation in exercises (severe chronic obstructive lung disease, severe heart failure, history of cerebrovascular events) 5-Hip and ankle problems 6-Participating in another physical therapy program in the last 3 months 7-History of intra-articular injections in the last 6 months

Ages: 45 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Visual Analog Scale (VAS) Change from baseline in pain on the VAS at month 3 | Baseline and month 3
  Visual Analog Scale (VAS) is used to measure and monitor the intensity of pain. This is a 10 cm ruler that describes painlessness at one end and the most severe pain at the other. A patient scores his/her pain from 0 to 10.

SECONDARY OUTCOMES:
Western OntarioMacMaster (WOMAC) Change from baseline in pain and physical functions on Western OntarioMacMaster scale at month | Baseline and month 3
  It is widely used in studies with knee OA patients. The scale, each question of which is evaluated with a 5-point Likert scale, consists of 24 questions. It is filled by patients. There are pain, physical function and stiffness subscales. Pain subscale is evaluated with five items and is scored between 0-20. The hardness subscale has two items and is scored between 0-8. Function subscale consists of 17 items and is scored between 0-68. A high score indicates poor function, pain or stiffness.
Femoral cartilage thickness Change from baseline in knee joint on the measuring the femoral cartilage thickness at month 3 | Baseline and month 3
  Femoral cartilage thickness is measured by the same physician by placing the probe axially in the suprapatellar region by ultrasonography while the patient is lying on his back and the knees are in maximum flexion. The distance between the thin hyperechoic line at the synovial cartilage interface and the sharp hyperechoic line at the cartilage-bone interface is defined as cartilage thickness

CONTACTS AND LOCATIONS:
Overall Officials: BANU ORDAHAN, Principal Investigator — Necmettin Erbakan University, Konya, Turkey
Locations (1):
- NEU, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No